CLINICAL TRIAL: NCT00017069
Title: CTI 1060: A Phase II Clinical Trial of Arsenic Trioxide and Dexamethasone as Therapy for Relapsed or Refractory Multiple Myeloma
Brief Title: Arsenic Trioxide and Dexamethasone in Treating Patients With Recurrent or Refractory Stage II or Stage III Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CTI-1060; CDR0000068646 (Registry Identifier: PDQ (Physician Data Query)); MSKCC-01012; NCI-G01-1951
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Arsenic Trioxide; Dexamethasone

INTERVENTIONS:
Drug: arsenic trioxide
Drug: dexamethasone

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combining arsenic trioxide and dexamethasone in treating patients who have recurrent or refractory stage II or stage III multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients with recurrent or refractory stage II or III multiple myeloma treated with arsenic trioxide and dexamethasone.
* Determine the rates of overall and relapse-free survival in patients treated with this regimen.
* Determine the safety profile of this treatment regimen in these patients.

OUTLINE: Patients receive arsenic trioxide IV daily for 5 days during the first week only and then 2 days a week thereafter. Patients also receive IV or oral dexamethasone on days 1-4 every 4 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity. Disease assessments are conducted every 4 weeks. Patients achieving complete response (CR) receive 2 additional courses of therapy after initial determination of CR.

Final assessments are conducted 4 weeks after the last study treatment and then annually thereafter.

PROJECTED ACCRUAL: A total of 55 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage II or III multiple myeloma
* Refractory myeloma defined as progressive disease (more than 25% increase in M protein or in radiographic findings of nonsecretory myeloma) despite up to 3 courses of prior cytotoxic chemotherapy

  * No more than 3 prior cytotoxic regimens
  * No more than 1 prior high-dose cytotoxic regimen with stem cell transplantation
* History of disease progression after prior steroid antimyeloma therapy
* No smoldering myeloma
* Measurable disease based on presence of serum and urine M protein and/or measurable plasmacytoma

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* Absolute granulocyte count greater than 1,200/mm^3*
* Platelet count greater than 75,000/mm^3*
* Hemoglobin greater than 10 g/dL* NOTE: *Unless due to multiple myeloma

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* SGOT and SGPT no greater than 2 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* Absolute QT interval less than 460 msec in the presence of normal potassium and magnesium levels
* No significant underlying cardiac dysfunction
* No conduction defects
* No unstable angina
* No congestive heart failure
* No New York Heart Association class II-IV cardiac disease
* No myocardial infarction within the past 6 months

Other:

* No preexisting grade 2 or greater neurotoxicity/neuropathy
* No other malignancy within the past 5 years except curatively treated carcinoma in situ of the cervix or nonmelanoma skin cancer
* No uncontrolled diabetes mellitus
* No active serious infection uncontrolled by antibiotics
* No history of grand mal seizures (other than infantile febrile seizures)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics
* See Chemotherapy
* At least 28 days since prior biologic therapy

Chemotherapy:

* See Disease Characteristics
* At least 28 days since prior cytotoxic chemotherapy, including high-dose cytotoxic regimen with stem cell transplantation
* No other concurrent cytotoxic chemotherapy

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* At least 28 days since prior radiotherapy except for focal radiation for symptom control

Surgery:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-02 (Actual); Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott C. Stromatt, MD, Study Chair — CTI BioPharma
Locations (10):
- United States (10):
  - Arizona Clinical Research Center, Tucson, Arizona
  - Highlands Oncology Group - Springdale, Springdale, Arkansas
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - Stockton Hematology Oncology Medical Group, Stockton, California
  - Rocky Mountain Cancer Centers - Midtown, Denver, Colorado
  - Pasco Pinellas Cancer Center - Tarpon Springs, Tarpon Springs, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Mountain States Tumor Institute - Boise, Meridian, Idaho
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Texas Cancer Care, Fort Worth, Texas